CLINICAL TRIAL: NCT01647308
Title: A Randomized, Double Blind, Placebo-Controlled, Phase 2 Study to Investigate the Effects of ISIS 304801 Lowering of ISIS-APOCIIIRX on Triglyceride Levels and Insulin Sensitivity in Subjects With Type 2 Diabetes Mellitus
Brief Title: Mechanistic Study of ISIS ISIS-APOCIIIRX in Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for business planning purposes. Assessments of APOCIIIRx in this population will be explored in a larger efficacy study
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 304801-CS4
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISIS-APOCIIIRX (Active Comparator)
  Interventions: Drug: ISIS-APOCIIIRX
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS-APOCIIIRX — 3 doses of ISIS ISIS-APOCIIIRX on alternate days during the first week and then once-weekly doses for 12 weeks.
  Arms: ISIS-APOCIIIRX
Drug: Placebo — 3 doses of placebo on alternate days during the first week and then once-weekly doses for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of ISIS ISIS-APOCIIIRX on Triglyceride Levels and Insulin Sensitivity in Subjects with Type 2 Diabetes on stable treatment with metformin.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 25 to </= 40 kg/m2
* Type 2 Diabetes Mellitus and on a stable dose of metformin
* Hypertriglyceridemia

Exclusion Criteria:

* Significant abnormalities in medical history, clinical examination or clinical testing
* Use of oral anti-diabetic medication other than metformin within 3 months prior to dosing
* History of outpatient insulin use for more than 2 weeks in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Total apoC-III | 91 Days
  The effect of treatment with ISIS ISIS-APOCIIIRX or Placebo on fasting total apoC-III levels.

SECONDARY OUTCOMES:
Insulin Sensitivity | Day 92
  Change from baseline in insulin sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States

REFERENCES:
- [Derived] Digenio A, Dunbar RL, Alexander VJ, Hompesch M, Morrow L, Lee RG, Graham MJ, Hughes SG, Yu R, Singleton W, Baker BF, Bhanot S, Crooke RM. Antisense-Mediated Lowering of Plasma Apolipoprotein C-III by Volanesorsen Improves Dyslipidemia and Insulin Sensitivity in Type 2 Diabetes. Diabetes Care. 2016 Aug;39(8):1408-15. doi: 10.2337/dc16-0126. Epub 2016 Jun 6. PMID 27271183